CLINICAL TRIAL: NCT06295432
Title: A Phase II, Multicenter Study to Assess the Safety, Tolerability and Anti-tumor Efficacy of DZD9008 in Combination With AZD4205 in Standard Treatment Failed Non-Small Cell Lung Cancer (NSCLC) Patients With EGFR Mutations
Brief Title: A Phase II Clinical Trial of DZD9008 in Combination With AZD4205 in Standard Treatment Failed NSCLC Patients With EGFR Mutations (WU-KONG21)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2022E0001
Record Dates: First submitted 2024-02-07; First posted 2024-03-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DZD9008+AZD4205 (Experimental): All subjects will receive both DZD9008 tablets and AZD4205 capsules orally. DZD9008 dosing will start at 200 mg daily, AZD4205 dosing will start at 75 mg daily.
  Interventions: Drug: DZD9008+AZD4205

INTERVENTIONS:
Drug: DZD9008+AZD4205 — Daily dose of DZD9008+AZD4205 until intolerant, disease progression or patient decision. Starting dose of DZD9008 is 200mg once daily and starting dose of AZD4205 is 75mg once daily orally used. If tolerated, subsequent cohorts will evaluate increasing doses of the combination therapy.
  Other Names: Inapplicable

SUMMARY:
DZD9008 in combination with AZD4205 for the treatment of patients with advanced NSCLC with EGFR mutations who have progressed after standard treatment. The purpose of this study is to assess the safety and efficacy of this combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the nature of the trial and provide a signed and dated informed consent form prior to screening.
2. Aged at least 18 years old when sign ICF.
3. Histological or cytological confirmed locally advanced or metastatic NSCLC.
4. Patients must exhibit Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1 at ICF signature with no deterioration over the previous 2 weeks.
5. Predicted life expectancy ≥ 12 weeks.
6. Patients with brain metastasis (BM) can only be enrolled under the condition that BM is previously treated and stable e.g. no evidence of progression for at least 2 weeks after CNS-directed treatment as ascertained by clinical examination and brain imaging (magnetic resonance image [MRI] or computed tomography [CT] scan) during the screening period), neurologically asymptomatic and not require corticosteroid treatment.
7. Adequate organ system functions, as outlined below

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Absolute lymphocyte count ≥ 0.8 x 109/L
   * Platelets ≥ 100 x 109/L
   * Hemoglobin ≥ 9 g/dL
   * Total bilirubin ≤ 1.5 x ULN if no liver metastases or ≤ 3 x ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN if no liver involvement or ≤ 5 x ULN with liver involvement
   * Creatinine ≤ 1.5 x ULN, or measured creatinine clearance ≥ 50 mL/min as calculated by the Cockcroft-Gault method
   * International normalized ratio (INR) ≤ 1.5 x ULN and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
   * Serum amylase ≤ 1.5 x ULN and serum lipase ≤ 1.5 x ULN
8. Male subjects with a female partner who intend to have children should use barrier contraception (e.g. condom) during their participation in the clinical study until 6 months after the last dose. Male subjects should not donate sperm during the clinical study until 6 months after the last dose. If the male subject has fertility requirements, it is recommended that sperm be frozen prior to the start of the clinical study.
9. Female subjects should use contraception at screening until 6 weeks after the last dose of DZD9008 or 3 months after the last dose of AZD4205, whichever is later, should not be breastfeeding and should have a negative pregnancy test (blood or urine β-HCG) at the time of screening.

Part A specific inclusion criteria:

1. Subjects should harbour any type of EGFR mutation.
2. Subjects should have progressed on, or be intolerant of prior standard systemic therapy for metastatic/locally advanced disease.

Part B specific inclusion criteria:

1. Subjects must have documented EGFR sensitizing mutation from a local certified laboratory.
2. Subjects should have progressed on, or be intolerant of prior standard systemic therapy for metastatic/locally advanced disease.
3. Patient must have measurable disease according to RECIST 1.1: At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for repeated measurement.
4. Agree and be willing to provide an adequate amount of the required tumor tissue for exploratory studies.

Exclusion Criteria:

1. Treatment with any of the followings:

   * Prior treatment with any onco-immunotherapy (e.g. PD-1) within 4 weeks before the first administration of IP.
   * Any cytotoxic chemotherapy, or other anticancer drugs from a previous treatment regimen within 2 weeks before the first administration of IP.
   * Radiotherapy within 2 weeks of the first dose or have not recovered from radiotherapy-related toxicity May receive palliative radiotherapy other than chest and brain, stereotactic radiosurgery and stereotactic body radiation therapy within 1 week prior to first dose a limited field of radiation for palliation within 1 week of the first administration of IP.
   * Patients currently receiving (or unable to stop using) medications known to be potent inhibitors or inducers of CYP3A or herbal supplements within 2 weeks before the first administration of IP.
   * Patients should avoid eating food known to be inhibitors of CYP3A such as grapefruit and Seville oranges (and other products containing these fruits, e.g., grapefruit juice or marmalade) within 2 weeks before the first administration of IP and 2 weeks after the therapy.
   * Drugs that prolong the QT interval need to be discontinued before the start of IP
   * Major surgery (excluding biopsy) within 4 weeks before the first administration of IP, or expect to have major surgery during study.
   * Treatment with any investigational drug (or unable to stop using) within 4 weeks before the first administration of IP
2. Spinal cord compression or leptomeningeal metastasis.
3. Prior malignancy within 2 years requires active treatment, except for adequately treated basal cell skin carcinoma, in situ cervical carcinoma, or other cancer type which has been disease free for > 2 years with life expectancy >2 years
4. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting IP with the exception of alopecia.
5. History of stroke or intracranial haemorrhage within 6 months before the first administration of IP.
6. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses (e.g., hemophilia, Von Willebrand disease).
7. Presence of persistent or active infection, including but not limited to:

   * Active or latent tuberculosis
   * Active herpes simplex, herpes zoster infection
   * COVID-19
   * active HBV, HCV, HIV infection
8. Any of the following cardiac abnormal and disease:

   * resting corrected QT interval (QTc) > 470 msec
   * Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block, and second-degree heart block, PR interval > 250 msec
   * Any factors that increase the risk of QTc prolongation, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
   * Prior history of atrial fibrillation except prior drug treatment related and recovered
   * Prior history of myocardial infarction, congestive heart failure, arrhythmias that are poorly controlled by medication
   * LVEF < 55% accessed by ECHO
9. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease, immunotherapy-induced immune pneumonitis.
10. Significant pulmonary function impairment (i.e. pulmonary function test showing FEV1 and DLCO < 60% of expected values).
11. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of IP.
12. Receiving live vaccines within 2 weeks before the first administration of IP.
13. Women who are pregnant or breast feeding.
14. Involvement in the planning and conduct of the study (applies to Dizal staff or staff at the study site).
15. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Part A: incidence of DLT , ≥grade 3 TEAEs and SAEs; Part B: incidence of ≥grade 3 TEAEs as assessed by CTCAE, incidence of SAEs. | DLT: 21 days after the first dose; AE that began after the start of trial medication treatment until 28 days after last dose.
  Part A: safety and tolerability of the combination therapy: incidence of DLT as defined in the protocol, incidence of ≥grade 3 TEAE as assessed by CTCAE, incidence of SAE; Part B: safety and tolerability of the combination therapy, to define RP2CD: incidence of ≥grade 3 TEAE as assessed by CTCAE, incidence of SAE.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, Principal Investigator — Guangdong Provincial People's Hospital
Locations (4):
- China (4):
  - Guangdong Provincial People'S Hospital, Guangzhou, Guangdong
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No